CLINICAL TRIAL: NCT02498236
Title: Target Engagement for Oxytocin: Response to 8 Doses
Brief Title: Target Engagement for Oxytocin: Dose Ranging Study
Acronym: R21Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Stephen R. Marder, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: R21
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia Spectrum
Keywords: Psychosis; Schizophrenia; Oxytocin
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin 6-84 IU (Experimental): Subjects will be randomly assigned to one of eight doses of intranasal oxytocin.
  Interventions: Drug: Intranasal Oxytocin
- Placebo (Placebo Comparator): Subjects will be administered intranasal placebo using the same spray volume as experimental condition
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin

SUMMARY:
This study will evaluate the effect of 8 doses of intranasal oxytocin or placebo on two proposed measures of target engagement in brain. The targets are (1) the suppression of a particular wave form (mu) on the electroencephalogram (EEG) while subjects observe a socially relevant form of motion and (2) pupil dilation will subjects identify faces showing different emotions.

DETAILED DESCRIPTION:
Subjects with schizophrenia spectrum disorders will be randomly assigned to one of 8 doses of oxytocin. After screening and informed consent subjects will receive either their assigned dose or a placebo. Thirty minutes following the drug administration patients will be evaluated on the EEG and pupillometry tasks followed by two tests that evaluate social salience. One week later subjects will have a second challenge in the alternative (drug or placebo) condition.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia, Schizoaffective Disorder, Delusional Disorder
* Able to cooperate with study procedures

Exclusion Criteria:

* Serious medical condition or substance use
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-09; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- 8IU Oxytocin: Subjects received either 8IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 12IU Oxytocin: Subjects received either 12IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 24IU Oxytocin: Subjects received either 24IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 36IU Oxytocin: Subjects received either 36IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 48IU Oxytocin: Subjects received either 48IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 60IU Oxytocin: Subjects received either 60IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 72IU Oxytocin: Subjects received either 72IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- 84IU Oxytocin: Subjects received either 84IU Oxytocin or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
Period: Overall Study
Arm/Group | 8IU Oxytocin | 12IU Oxytocin | 24IU Oxytocin | 36IU Oxytocin | 48IU Oxytocin | 60IU Oxytocin | 72IU Oxytocin | 84IU Oxytocin
Started | 6 | 6 | 6 | 6 | 7 | 6 | 7 | 7
Randomized | 6 | 6 | 6 | 6 | 7 | 6 | 7 | 7
Completed | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Did not show for testing | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Equipment failure | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed both study visits
Groups:
- 8IU Oxytocin; 12IU Oxytocin; 24IU Oxytocin; 36IU Oxytocin; 48IU Oxytocin; 60IU Oxytocin; 72IU Oxytocin; 84IU Oxytocin: Subjects received either the assigned Oxytocin dose or placebo 30 minutes prior to study assessments, and a second challenge in the alternative (drug or placebo) condition one week later.
- Total: Total of all reporting groups
Arm/Group | 8IU Oxytocin | 12IU Oxytocin | 24IU Oxytocin | 36IU Oxytocin | 48IU Oxytocin | 60IU Oxytocin | 72IU Oxytocin | 84IU Oxytocin | Total
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (8.1) | 45.3 (9.2) | 42.2 (11.9) | 45.5 (8.7) | 43.3 (10.0) | 45.2 (9.8) | 37.2 (11.3) | 43.0 (9.8) | 42.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each row corresponds to a dose of oxytocin. The sum of the participants in each row totals 47, which is the overall analyzed population.
  Participants
    Female | 2 | 3 | 2 | 2 | 3 | 1 | 1 | 2 | 16
    Male | 3 | 3 | 4 | 4 | 3 | 5 | 5 | 4 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row corresponds to a dose of oxytocin. The sum of the participants in each row totals 47, which is the overall analyzed population.
  Participants
    Hispanic or Latino | 1 | 3 | 1 | 0 | 1 | 1 | 2 | 1 | 10
    Not Hispanic or Latino | 4 | 3 | 5 | 6 | 5 | 5 | 4 | 5 | 37
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row corresponds to a dose of oxytocin. The sum of the participants in each row totals 47, which is the overall analyzed population.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 3 | 1 | 2 | 5 | 1 | 2 | 3 | 2 | 19
    White | 1 | 4 | 3 | 1 | 4 | 4 | 2 | 4 | 23
    More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 47

OUTCOME MEASURES:

1. Primary Outcome: Mu Suppression on EEG
Description: This primary outcome measure is mu suppression recorded during a biological motion task. In this task, participants view point-light walker (PLW) animations of a human; the PLWs were either male or female, happy or sad, or walking towards or away from the viewer. In addition to the humans, there was a control condition which consisted of a circle moving either left or right. In separate blocks, participants had to identify either the gender, the emotion, or intention (i.e., direction) of the walker, or the direction of the circle, while their EEG was recorded. The primary measure was mu activity (8-12 Hz) recorded over 3 central electrodes. Mu suppression was calculated as the log10 transformed ratio of mu power to one of the three human conditions compared to the circle: log10(human/circle). A negative value indicates suppression of mu activity to human walkers vs. circles. We are presenting the mean (SD) of this suppression ratio collapsed over the 3 human conditions.
Time Frame: Baseline, 1 Week
Measure: Mean (Standard Deviation); unit: log10 transformed ratio (Hz)
Groups:
- 8IU Oxytocin: 8 international units (IU) of Oxytocin
- 12IU Oxytocin: 12 international units (IU) of Oxytocin
- 24IU Oxytocin: 24 international units (IU) of Oxytocin
- 36IU Oxytocin: 36 international units (IU) of Oxytocin
- 48IU Oxytocin: 48 international units (IU) of Oxytocin
- 60IU Oxytocin: 60 international units (IU) of Oxytocin
- 72IU Oxytocin: 72 international units (IU) of Oxytocin
- 84IU Oxytocin: 84 international units (IU) of Oxytocin
- Placebo: Placebo condition. This represents the placebo data summarized across all participants regardless as to which dose of oxytocin (OT) they received.
Arm/Group | 8IU Oxytocin | 12IU Oxytocin | 24IU Oxytocin | 36IU Oxytocin | 48IU Oxytocin | 60IU Oxytocin | 72IU Oxytocin | 84IU Oxytocin | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 47
log10 transformed ratio (Hz) | -0.0907 (0.10515) | -0.0632 (0.08206) | -0.0542 (0.07471) | -0.1153 (0.07699) | -0.1333 (0.06625) | -0.0459 (0.03514) | -0.1101 (0.02654) | -0.0149 (0.08074) | -0.0726 (0.10331)

2. Primary Outcome: Pupil Dilation While Observing Faces
Description: This primary outcome measure is pupil size recorded during a facial affect identification task. In this task, participants view faces portraying happy, afraid, or neutral faces; scrambled images of the faces were also shown. There were 64 trials: 16 trials per each image type. The primary measure was the difference in pupil size averaged over the happy and fearful faces from the scrambled face condition. A positive value indicates greater pupil dilation relative to the scrambled face; a negative value indicates greater pupil constriction relative to the scrambled face.
  Baseline was defined as the median pupil width 1 second prior to stimulus onset. Pupil sizes during each trial were baseline-corrected by dividing them by baseline median width. Resulting pupil size timecourses were averaged within-subject for each type of stimulus (happy, afraid, neutral, scrambled). The primary dependent variable was computed by taking the average of the change in pupil size between 1 and 3 s.
Time Frame: Baseline, 1 Week
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Placebo: Placebo condition. This represents the placebo data summarized across all participants regardless as to which dose of OT they received.
Arm/Group | 8IU Oxytocin | 12IU Oxytocin | 24IU Oxytocin | 36IU Oxytocin | 48IU Oxytocin | 60IU Oxytocin | 72IU Oxytocin | 84IU Oxytocin | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 47
arbitrary units | .0074 (.00669) | .0347 (.03395) | -.0089 (04525) | .0153 (.02317) | -.0011 (.02862) | .0103 (.01498) | .0299 (.03634) | .0073 (.03469) | .0134 (.03195)

ADVERSE EVENTS:
Time Frame: One week. Participants were only enrolled for a one week period in which placebo or drug were administered (in random order) either at baseline or 1-week follow-up.
Arm/Group | 8IU Oxytocin | 12IU Oxytocin | 24IU Oxytocin | 36IU Oxytocin | 48IU Oxytocin | 60IU Oxytocin | 72IU Oxytocin | 84IU Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/47
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT02498236/Prot_SAP_ICF_000.pdf